CLINICAL TRIAL: NCT04852835
Title: Follow-up of COVID-19 Vaccine Response in Strasbourg University Hospitals
Acronym: COVACHUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8223
Record Dates: First submitted 2021-04-07; First posted 2021-04-21 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 Vaccines
Keywords: COVID-19; SARS-CoV-2; Vaccine; Humoral response; Anti-spike antibodies; Neutralizing antibodies; Gender
MeSH Terms: conditions — COVID-19; Coitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vaccination remains the main promising measure to fight against the COVID-19 pandemic. The presumed efficacy of the vaccines is quite remarkable since it varies between 62 and 95%. There is increasing evidence that sex-specific effects may lead to different outcomes of vaccine safety and efficacy. However, sex-disaggregated data after COVID-19 vaccine are lacking. The first purpose of the study is to determine antibody titers against SARS-CoV-2 spike after COVID-19 vaccination. The secondary purpose is to identify predictor factors of immune response including age, gender and biological factors.

ELIGIBILITY:
Inclusion Criteria:

- Any person, male or female, over 18 years of age who underwent vaccination and

* anti-SARS-CoV-2 serological test after vaccination
* having already given their consent for their biological resources to be:

  * stored in a biocollection of the Microbiology Technical Platform (PTM) having received an approval from the CPP Est-IV and declared to the Ministry of Education and Research under reference No. DC2009-1002;
  * subsequently reused, as well as the anonymized associated data, for research purposes

Exclusion Criteria:

* Inability to give clear information (person in an emergency, difficulty understanding the subject, etc.)
* Person under safeguard of justice
* Person under guardianship or curatorship-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any person, male or female, over 18 years of age who underwent vaccination and anti-SARS-CoV-2 serological test after vaccination
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Study of the relationship between the serological response to the COVID-19 vaccine and the demographic characteristics of the patient | up to 1 month post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Samira FAFI-KREMER, PharmD, PhD, Study Director — Service de Virologie - Hôpital Civil
Locations (1):
- Service de Virologie - Hôpital Civil, Strasbourg, France